CLINICAL TRIAL: NCT03072992
Title: Study of Efficacy of Curcumin in Combination With Chemotherapy in Patients With Advanced Breast Cancer: Randomized, Double Blind, Placebo Controlled Clinical Trial
Brief Title: "Curcumin" in Combination With Chemotherapy in Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center of Oncology, Armenia (Other)
Collaborators: BRIU GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5592-17-02-23
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Curcumin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Paclitaxel & Curcumin (Active Comparator): 75 patients, treatment with Curcumin (CUC-01, yellow solution), 300mg i.v. plus i.v. Paclitaxel (colorless solution) 80 mg /m2 BS i.e., once weekly for 12 weeks.
  Interventions: Drug: Curcumin; Drug: Paclitaxel
- Group B: Paclitaxel & Placebo (Placebo Comparator): Group B, 75 patients, treatment with Paclitaxel (colorless solution) 80 mg /m2 BS, i.v. plus placebo i.v. solution (250 ml, yellow solution for masking/blinding), once weekly for 12 weeks.
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Curcumin — Curcumin (CUC-01), 300mg i.v. , once weekly for 12 weeks.
  Other Names: CUC-01
  Arms: Group A: Paclitaxel & Curcumin
Drug: Paclitaxel — Paclitaxel (colorless solution) 80 mg /m2 BS, i.v., once weekly for 12 weeks.
Drug: Placebo — Placebo i.v. solution, once weekly for 12 weeks
  Arms: Group B: Paclitaxel & Placebo

SUMMARY:
The aim of this study is to assess benefits of treatment with intravenous Curcumin® (CUC-01) vs placebo, in combination with paclitaxel chemotherapy, and to estimate the risk of adverse events in patients with locally advanced and metastatic breast cancer.

This is a randomized, double-blind, placebo-controlled, two arms parallel group phase 2 clinical trial:

Group A, 75 patients, treatment with Curcumin (CUC-01, yellow solution), 300mg i.v. plus i.v. Paclitaxel (colorless solution) 80 mg /m2 BS i.e., once weekly for 12 weeks.

Group B, 75 patients, treatment with Paclitaxel (colorless solution) 80 mg /m2 BS, i.v. plus placebo i.v. solution (250 ml, yellow solution for masking/blinding), once weekly for 12 weeks.

Primary objective of the study:

To assess:

* Efficacy of combined therapy with Curcumin ®, (CUC-01) and Paclitaxel vs Paclitaxel in patients with advanced and metastatic breast cancer in terms of Objective Response Rate (ORR) assessed with the Modified Response Evaluation Criteria In Solid Tumours (RECIST).

Secondary objectives of the study:

To assess:

* The safety of Curcumin+Paclitaxel combination compared to Paclitaxel+placebo treatment by assessment of adverse effects.
* Quality of life (QOL) in patient treated with Curcumin+Paclitaxel combination compared to Paclitaxel+Placebo
* Response duration in terms of Progression free survival (PFS), Time to Disease Progression (TTP) and Time to treatment failure (TTTF)

DETAILED DESCRIPTION:
RATIONALE

Various preclinical, clinical, and animal studies suggest that curcumin has potential as an antiproliferative, anti-invasive, and antiangiogenic, as a mediator of chemoresistance, chemopreventive, and as a therapeutic agent. However, the main problem associated with the use of curcumin in humans is its low absorption from the gastrointestinal tract, poor solubility in body fluids and low bioavailability. To overcome the pharmacokinetic and bioavailability limitations of oral administration, water soluble curcumin, Curcumin® (CUC-01) injection, a clear, yellow viscous solution intended for dilution with a suitable parenteral fluid prior to intravenous infusion was elaborated. Curcumin® (CUC-01) injection is patented pharmacy product and sold per individual prescription in Germany and other countries for Cancer Centers. However, clinical efficacy and safety of these formulation have to be confirmed in this study.

Development of multidrug resistance (MDR) against a variety of conventional and novel chemotherapeutic agents is a significant challenge in effective cancer therapy. Paclitaxel, one of the most prescribed conventional chemotherapeutic agents, acts as microtubule stabilizer and blocks cancer cells in the G2/M phase, thus preventing them from mitosis. It is also an apoptosis inducer in cancer cells. However, one of the main drawbacks of its use is that it is also a substrate of P-gp and treatment with PCL induces the overexpression of the efflux pump in the cancer cells. NF-κB is a transcription factor that controls the expression of genes involved in a number of physiological responses including differentiation, inflammation, apoptosis and upregulation of the P-gp. The PI3K/Akt pathway is also another over-activated pathway in a wide range of tumor types and therefore its over-activation leads to increased cancer-cell survival, proliferation, and growth and it also promotes NF-κB activity, all affects the success of the chemotherapy with Paclitaxel. Curcumin is known to downregulate both the PI3K/Akt and NF-κB pathways independent of each other, and thus it can act as a mediator of chemoresistance by sensitizing cancer cells to a conventional chemotherapeutic agents.

It has been suggested that co-administration of Paclitaxel and curcumin will help to overcome multidrug resistance in cancer. Synergistic interaction of curcumin and paclitaxel was demonstrated in paclitaxel (Taxol)-resistant breast cancer cells, human breast cancer xenograft model, in MDA-MB-231 and MCF-7 human breast cancer cells and many other cancer cell lines. In vivo, this combination treatment produced a three-fold tumor inhibition with each of these cell lines. Furthermore, the combination of paclitaxel and curcumin exerted increased anti-tumor efficacy on mouse models These results clearly indicate combination of Curcumin with paclitaxel could have significant clinical advantages for the treatment of breast cancer.

Curcumin exerted in vitro anti-breast cancer activities through regulation of matrix metalloproteinase (MMP)-2, B-cell lymphoma 2 (Bcl-2), Bax, flap endonuclease 1 (Fen1), NF-E2-related factor 2 (Nrf-2) factors, and phosphoinositide 3-kinase (PI3K)/protein kinase B (Akt) signaling.

Therefore, and based on this evaluation, we intend examining the effect of Curcumin ®, (CUC-01) in advanced and metastatic breast cancer in this randomized, double-blind, placebo-controlled study.

STUDY DESIGN

This is a randomized, double-blind, placebo-controlled, two arms parallel group phase 2 study:

Group A, 75 patients, treatment with Curcumin (CUC-01, yellow solution), 300mg i.v. plus i.v. Paclitaxel (colorless solution) 80 mg /m2 BS i.e., once weekly for 12 weeks.

Group B, 75 patients, treatment with Paclitaxel (colorless solution) 80 mg /m2 BS, i.v. plus placebo i.v. solution (250 ml, yellow solution for masking/blinding), once weekly for 12 weeks.

Therapy schedule weekly:

* Preload-infusion containing Dexamethasone 8 mg in 100ml NaCl
* Paclitaxel 80mg/m2 body surface in 250 ml 0.9% NaCl
* Curcumin 300 mg or placebo in 250ml 0.9% NaCl

PRIMARY OBJECTIVE

To assess:

* Efficacy of combined therapy with Curcumin ®, (CUC-01) and Paclitaxel vs Paclitaxel in patients with advanced and metastatic breast cancer in terms of Objective Response Rate (ORR)

SECONDARY OBJECTIVES

To assess:

* The safety of Curcumin+Paclitaxel combination compared to Paclitaxel+placebo treatment by assessment of adverse effects.
* Quality of life (QOL) in patient treated with Curcumin+Paclitaxel combination compared to Paclitaxel+Placebo
* Response duration in terms of Progression free survival (PFS), and Time to Disease Progression (TTP) and Time to treatment failure (TTTF)

NUMBER OF SUBJECTS

150

TEST PRODUCT, DOSE, AND ROUTE OF ADMINISTRATION

Curcumin® (CUC-01) injection, BRIU GmbH at dose 300 mg. Each vial contains 20 ml of the concentrate (concentration of Curcumin - 15 mg/ml) containing in total of 300 mg of Curcumin, which has to be diluted in 250 ml of physiological solution (0.9% NaCl) before use, total volume - 270 ml of infusion solution.

Investigational Active Ingredients: Curcuminoids (syn: Curcumin, isolated from turmeric rhizome Curcuma longa, Zingiberaceae.

CUC-01 will be administered intravenously (IV) once in every 7 days for 12 weeks.

Therapy schedule weekly:

* Preload-infusion containing Dexamethasone 8 mg in 100ml NaCl
* Curcumin 300 mg in 250ml 0.9% NaCl
* Paclitaxel 80mg/m2 body surface in 250 ml o.9% NaCl

CONTROL PRODUCT, DOSE AND ROUTE OF ADMINISTRATION

Placebo: Riboflavin solution which has strong yellow-orange color and visually is not distinguishable from Curcumin.

Placebo will be administered intravenously (IV) once in every 7 days for 12 weeks

Therapy schedule weekly:

* Preload-infusion containing Dexamethasone 8 mg in 100ml NaCl
* Placebo(Riboflavin solution) in 250ml 0,9% NaCl
* Paclitaxel 80mg/m2 body surface in 250 ml 0.9% NaCl

EFFICACY EVALUATIONS.

Primary endpoint

Primary outcome measures:

Clinically, radiologically measurable disease, tumour markers:

* Objective response rate, assessed with the Modified Response Evaluation Criteria In Solid Tumours (RECIST) using plain radiographs, ultrasound imaging, computed tomography scans and magnetic resonance imaging. Other studies may be acceptable with the approval of the principal investigator.
* Carcinoembryonic antigen (CEA) assay and Cancer antigen15-3 (CA 15-3) assay

Secondary endpoints.

Secondary outcome measures:

* Adverse events and defined by National Cancer Institute (NCI) Common Toxicity Criteria Version 4.0 (CTCAE, v4.0≤)
* Quality of Life measures (EORTC QLQ-C30, Global Health Status/QoL scales)Response Duration measures:
* Progression free survival (PFS) assessed from study enrolment to tumour progression as per the Modified RECIST criteria or disease related
* Time to Treatment Failure (TTTF), assessed from study enrolment to cessation of study treatment for any reason
* Time to Tumour Progression (TTP), assessed from study enrolment to tumour progression as per the Modified RECIST criteria.

Safety Evaluations

Tolerability will be assessed by the nature and incidence of adverse events. Change in clinical safety labs from baseline to end of the study Incidence of adverse events, (CTCAE, v4.0≤).

STATISTICS

Statistical analysis will be performed on an intent-to-treat basis. Survival Analysis for time-to event endpoints.

Assessment of baseline characteristics - between groups comparison will be made by:

* Kruskal-Wallis (KW) non-parametric one way ANOVA rank order test, with post hoc Dunn's Multiple Comparison Test or
* parametric One-way independent measures ANOVA with Dunnett's Multiple Comparison Test,

Analysis of changes within treatment groups in the course of the study (before versus after) was performed by:

* paired t-test (parametric data - variables with normal distribution) or/and
* Wilcoxon signed rink test (nonparametric data), or
* Friedman test for repeated several measures (nonparametric data),

Assessment of efficacy of study medications was achieved by between groups comparison of mean changes from the baseline (differences before and after treatment of every single patient) using:

* Kruskal-Wallis (KW) non-parametric one way ANOVA rank order test, with post hoc Dunn's Multiple Comparison Test, and/or
* parametric One-way independent measures ANOVA with Tukkey's Multiple Comparison Test (variables with normal distribution).

Survival Analysis Statistical tools (Kaplan-Mayer analysis with log-rank test, Cox regression etc.) will be used for assessment of the TTP, PFS and TTTF.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients must fulfill all the following criteria to be eligible for this study.
* Patient should be able to give fully informed written consent according to International Conference on Harmonisation (ICH)/Good Clinical Practice (GCP) guidelines and to comply with the instructions in the protocol.
* Patients should be diagnosed with histologically-proven breast carcinoma.
* Female subjects 18 years or older.
* Radiographic evidence of measurable disease is required and must have been performed within 8 weeks prior to randomization. Acceptable studies include plain radiographs, ultrasound imaging, computed tomography scans and magnetic resonance imaging. Other studies may be acceptable with the approval of the principal investigator.
* Bidimensionally measurable manifestations of progressive advanced disease after one prior chemotherapy regimen, or locally advanced or MBC that progressed during or within 12 months of completing an adjuvant or neoadjuvant chemotherapy regimen or other cases of breast cancer in which weekly paclitaxel treatment is considered an adequate approach.
* No Herceptin treatment 4 weeks before and during the study.
* No other chemotherapy and bisphosphonate therapy 4 weeks before random assignment and during the study. Prior and concomitant hormonal therapy is allowed.
* Karnofsky performance score (KPS) ≥60, ECOG≤2.
* Life expectancy 3 month or greater, as estimated by the responsible clinician.
* Women of child-bearing age must use effective contraception.
* Sufficient hematological status. Adequate bone marrow function defined as:

  * WBC greater than 4.0 x 10^9/L
  * Granulocyte count greater than 1.5 x 10^9/L
  * Platelet count greater than 100 x 10^9/L
  * Haemoglobin greater than 10 g/dl;
* Adequate renal function: calculated creatinine clearance (Cockcroft-Gault formula) greater than 45 ml/min;
* Adequate hepatic function defined as a total bilirubin less than Upper Limit of Normal (ULN), Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) less than 2.5 x ULN, or 1.5 x ULN if Alkaline Phosphatase (Alk Phos) less than 2.5 x ULN. Alk Phos less than 5 x ULN unless patient has bone metastases;

EXCLUSION CRITERIA:

* inadequate renal and hepatic functions;
* inadequate haematological status;
* uncontrolled central nervous system metastases;
* severe cardiovascular disorders;
* active infection;
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements;
* Other non-malignant systemic and/or other disease, that would preclude the patient from receiving study treatment or would prevent required follow-up (at the discretion of the principal investigator);
* Known hypersensitivity to any of the study drugs or excipients;
* Pregnancy or lactation;
* Second primary malignancy diagnosed within the last 5 years (except for adequately treated non-melanoma skin cancers and in-situ cervical carcinoma adequately treated by cone excision);
* Herceptin and/or chemotherapy and/or bisphosphonate therapy less than 4 weeks before the randomisation;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 4 weeks after the completion of the treatment
  Objective response rate, assessed with the Modified Response Evaluation Criteria In Solid Tumours (RECIST).

SECONDARY OUTCOMES:
Adverse events | 24 weeks
  Adverse events and defined by National Cancer Institute (NCI) Common Toxicity Criteria Version 4.0 (CTCAE, v4.0≤).
Global Health Status/QoL scale | 24 weeks
  Health status measured by Global Health Status/QoL scale of EORTC QLQ-C30.
Progression free survival | 24 weeks
  Progression free survival assessed from study enrolment to tumour progression as per the Modified RECIST criteria.
Time to Treatment Failure | 24 weeks
  Time to Treatment Failure assessed from study enrolment to cessation of study treatment for any reason.
Time to Tumour Progression | 24 weeks
  Time to Tumour Progression assessed from study enrolment to tumour progression as per the Modified RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Armen Tananyan, PhD, Study Chair — National Center of Oncology, Armenia
Locations (1):
- National Center of Oncology, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: Undecided